CLINICAL TRIAL: NCT02653742
Title: Prospective, Randomized, Allocation-Concealed, Blinded Study Designed to Compare Ketorolac Sublingual and Fentanyl Intranasal in Pain Control for Bilateral Myringotomy and Tubes (BMT) Placement in Children
Brief Title: Ketorolac Sublingual vs. Fentanyl Intranasal in Pain Control for Bilateral Myringotomy and Tubes (BMT) Placement in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anica Crnkovic (Other)
Responsible Party: Sponsor-Investigator, Anica Crnkovic, Anesthesiologist, Albany Medical College
Organization: Albany Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3943
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Pain, Postoperative; Otitis Media
MeSH Terms: conditions — Pain, Postoperative; Otitis Media | interventions — Ketorolac; Ketorolac Tromethamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (3):
- Ketorolac (Experimental): Ketorolac 1mg/kg sublingual, in the form of Ketorolac Tromethamine solution for intravenous/intramuscular use.
  Interventions: Drug: Ketorolac
- Fentanyl (Experimental): Fentanyl 2mcg/kg intranasal, in the form of Fentanyl Citrate solution for intravenous/intramuscular use.
  Interventions: Drug: Fentanyl
- Ketorolac and Fentanyl (Experimental): Ketorolac 1mg/kg sublingual, in the form of Ketorolac Tromethamine solution for intravenous/intramuscular use and Fentanyl 2mcg/kg intranasal, in the form of Fentanyl Citrate solution for intravenous/intramuscular use.
  Interventions: Drug: Ketorolac; Drug: Fentanyl

INTERVENTIONS:
Drug: Ketorolac — Ketorolac 1mg/kg sublingual is administered after induction of general anesthesia.
  Other Names: Toradol
  Arms: Ketorolac; Ketorolac and Fentanyl
Drug: Fentanyl — Fentanyl 2mg/kg intranasal is administered after induction of general anesthesia
  Arms: Fentanyl; Ketorolac and Fentanyl

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ketorolac sublingual with fentanyl intranasal used in our hospital for pain control in children undergoing bilateral myringotomy with placement of pressure equalization tubes (BMTs).

DETAILED DESCRIPTION:
This prospective, randomized, allocation concealed blinded study is designed to compare ketorolac sublingual vs. fentanyl intranasal vs. the combination of these two medications for pain control after BMTs in children. Bilateral myringotomy and tube placement is an elective operation, mainly in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) I-II physical class
* Scheduled for elective BMT
* Mask induction of anesthesia

Exclusion Criteria:

* Allergy to any NSAIDs
* Severe upper respirator infection
* Severe asthma
* Bleeding disorders
* History of GI bleeding
* Renal impairment
* Scheduled for one-sided myringotomy and tube placement

Ages: 8 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain score assessment | Through study completion, an average of 1 hour postop
  Pain assessment score using CHEOPS

SECONDARY OUTCOMES:
Administration of additional pain medication | Through study completion, an average of 1 hour postop
  The need for additional pain medication other than the study medication to control postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Anica Crnkovic, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

REFERENCES:
- [Background] Croteau N, Hai V, Pless IB, Infante-Rivard C. Trends in medical visits and surgery for otitis media among children. Am J Dis Child. 1990 May;144(5):535-8. doi: 10.1001/archpedi.1990.02150290029019. PMID 2330920
- [Background] Watcha MF, Ramirez-Ruiz M, White PF, Jones MB, Lagueruela RG, Terkonda RP. Perioperative effects of oral ketorolac and acetaminophen in children undergoing bilateral myringotomy. Can J Anaesth. 1992 Sep;39(7):649-54. doi: 10.1007/BF03008224. PMID 1394752
- [Background] Aldrete JA, Kroulik D. A postanesthetic recovery score. Anesth Analg. 1970 Nov-Dec;49(6):924-34. No abstract available. PMID 5534693
- [Background] Moodie JE, Brown CR, Bisley EJ, Weber HU, Bynum L. The safety and analgesic efficacy of intranasal ketorolac in patients with postoperative pain. Anesth Analg. 2008 Dec;107(6):2025-31. doi: 10.1213/ane.0b013e318188b736. PMID 19020154
- [Background] Gupta A, Daggett C, Ludwick J, Wells W, Lewis A. Ketorolac after congenital heart surgery: does it increase the risk of significant bleeding complications? Paediatr Anaesth. 2005 Feb;15(2):139-42. doi: 10.1111/j.1460-9592.2005.01409.x. PMID 15675931
- [Background] Aldrink JH, Ma M, Wang W, Caniano DA, Wispe J, Puthoff T. Safety of ketorolac in surgical neonates and infants 0 to 3 months old. J Pediatr Surg. 2011 Jun;46(6):1081-5. doi: 10.1016/j.jpedsurg.2011.03.031. PMID 21683202
- [Background] Papacci P, De Francisci G, Iacobucci T, Giannantonio C, De Carolis MP, Zecca E, Romagnoli C. Use of intravenous ketorolac in the neonate and premature babies. Paediatr Anaesth. 2004 Jun;14(6):487-92. doi: 10.1111/j.1460-9592.2004.01250.x. PMID 15153212
- [Background] Lynn AM, Bradford H, Kantor ED, Andrew M, Vicini P, Anderson GD. Ketorolac tromethamine: stereo-specific pharmacokinetics and single-dose use in postoperative infants aged 2-6 months. Paediatr Anaesth. 2011 Mar;21(3):325-34. doi: 10.1111/j.1460-9592.2010.03484.x. Epub 2010 Dec 29. PMID 21199130
- [Background] Cohen MN, Christians U, Henthorn T, Vu Tran Z, Moll V, Zuk J, Galinkin J. Pharmacokinetics of single-dose intravenous ketorolac in infants aged 2-11 months. Anesth Analg. 2011 Mar;112(3):655-60. doi: 10.1213/ANE.0b013e3182075d04. Epub 2011 Jan 13. PMID 21233498
- [Background] Pappas AL, Fluder EM, Creech S, Hotaling A, Park A. Postoperative analgesia in children undergoing myringotomy and placement equalization tubes in ambulatory surgery. Anesth Analg. 2003 Jun;96(6):1621-1624. doi: 10.1213/01.ANE.0000064206.51296.1D. PMID 12760984
- [Background] Zuppa AF, Mondick JT, Davis L, Cohen D. Population pharmacokinetics of ketorolac in neonates and young infants. Am J Ther. 2009 Mar-Apr;16(2):143-6. doi: 10.1097/MJT.0b013e31818071df. PMID 19300040
- [Background] Neri E, Maestro A, Minen F, Montico M, Ronfani L, Zanon D, Favret A, Messi G, Barbi E. Sublingual ketorolac versus sublingual tramadol for moderate to severe post-traumatic bone pain in children: a double-blind, randomised, controlled trial. Arch Dis Child. 2013 Sep;98(9):721-4. doi: 10.1136/archdischild-2012-303527. Epub 2013 May 23. PMID 23702435
- [Background] Gupta A, Daggett C, Drant S, Rivero N, Lewis A. Prospective randomized trial of ketorolac after congenital heart surgery. J Cardiothorac Vasc Anesth. 2004 Aug;18(4):454-7. doi: 10.1053/j.jvca.2004.05.024. PMID 15365927
- [Background] Perez-Urizar J, Aguilar-Cota ME, Herrera JE, Flores-Murrieta FJ. Comparative bioavailability of ketorolac tromethamine after intramuscular and sublingual administration. Proc West Pharmacol Soc. 2002;45:6-7. No abstract available. PMID 12434509
- [Background] Drover DR, Hammer GB, Anderson BJ. The pharmacokinetics of ketorolac after single postoperative intranasal administration in adolescent patients. Anesth Analg. 2012 Jun;114(6):1270-6. doi: 10.1213/ANE.0b013e31824f92c2. Epub 2012 Mar 30. PMID 22467894
- [Background] He A, Hersh EV. A review of intranasal ketorolac tromethamine for the short-term management of moderate to moderately severe pain that requires analgesia at the opioid level. Curr Med Res Opin. 2012 Dec;28(12):1873-80. doi: 10.1185/03007995.2012.744302. Epub 2012 Nov 9. PMID 23098098
- [Background] Garnock-Jones KP. Intranasal ketorolac: for short-term pain management. Clin Drug Investig. 2012 Jun 1;32(6):361-71. doi: 10.2165/11209240-000000000-00000. PMID 22574632
- [Background] Finkel JC, Cohen IT, Hannallah RS, Patel KM, Kim MS, Hummer KA, Choi SS, Pena M, Schreiber SB, Zalzal G. The effect of intranasal fentanyl on the emergence characteristics after sevoflurane anesthesia in children undergoing surgery for bilateral myringotomy tube placement. Anesth Analg. 2001 May;92(5):1164-8. doi: 10.1097/00000539-200105000-00016. PMID 11323340
- [Background] Galinkin JL, Fazi LM, Cuy RM, Chiavacci RM, Kurth CD, Shah UK, Jacobs IN, Watcha MF. Use of intranasal fentanyl in children undergoing myringotomy and tube placement during halothane and sevoflurane anesthesia. Anesthesiology. 2000 Dec;93(6):1378-83. doi: 10.1097/00000542-200012000-00006. PMID 11149429
- [Background] Karl HW, Rosenberger JL, Larach MG, Ruffle JM. Transmucosal administration of midazolam for premedication of pediatric patients. Comparison of the nasal and sublingual routes. Anesthesiology. 1993 May;78(5):885-91. doi: 10.1097/00000542-199305000-00013. PMID 8489062
- [Background] Bean-Lijewski JD, Stinson JC. Acetaminophen or ketorolac for post myringotomy pain in children? A prospective, double-blinded comparison. Paediatr Anaesth. 1997;7(2):131-7. doi: 10.1046/j.1460-9592.1997.d01-47.x. PMID 9188114
- [Background] Forrest JB, Heitlinger EL, Revell S. Ketorolac for postoperative pain management in children. Drug Saf. 1997 May;16(5):309-29. doi: 10.2165/00002018-199716050-00003. PMID 9187531
- [Background] Davis PJ, Greenberg JA, Gendelman M, Fertal K. Recovery characteristics of sevoflurane and halothane in preschool-aged children undergoing bilateral myringotomy and pressure equalization tube insertion. Anesth Analg. 1999 Jan;88(1):34-8. doi: 10.1097/00000539-199901000-00007. PMID 9895062
- [Background] Lynn AM, Bradford H, Kantor ED, Seng KY, Salinger DH, Chen J, Ellenbogen RG, Vicini P, Anderson GD. Postoperative ketorolac tromethamine use in infants aged 6-18 months: the effect on morphine usage, safety assessment, and stereo-specific pharmacokinetics. Anesth Analg. 2007 May;104(5):1040-51, tables of contents. doi: 10.1213/01.ane.0000260320.60867.6c. PMID 17456651